CLINICAL TRIAL: NCT07332000
Title: A Biomarker Study in Men With Localized Prostate Cancer Treated With Aglatimagene Besadenovec
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PrTK05
Record Dates: First submitted 2025-12-17; First posted 2026-01-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer Patients Treated by Radiotherapy
Keywords: Biomarkers; Viral Shedding
MeSH Terms: interventions — Valacyclovir; Prodrugs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients receiving the experimental drug
  Interventions: Biological: aglatimagene besadenovec + valacyclovir

INTERVENTIONS:
Biological: aglatimagene besadenovec + valacyclovir — This is an open-label, single-group study in which up to 30 participants diagnosed with localized favorable intermediate-risk prostate cancer, with planned external beam radiation therapy (EBRT) treatment, will receive 3 intraprostatic injections of aglatimagene besadenovec each, followed by 14-day courses of valacyclovir. Participants will have aglatimagene besadenovec administered either transrectally or transperineally.
  Other Names: CAN-2409 plus prodrug

SUMMARY:
Phase 2a, open-label, multi-center study evaluating biomarkers and biodistribution of aglatimagene besadenovec plus valacyclovir in men with localized, favorable intermediate-risk prostate cancer who are planning to receive external beam radiation therapy (EBRT).

DETAILED DESCRIPTION:
This is a phase 2a, open-label, multi-center study evaluating aglatimagene besadenovec plus prodrug in men with localized, favorable intermediate-risk prostate cancer who are planning to receive external beam radiation therapy (EBRT). Aglatimagene besadenovec is a replication-deficient adenoviral vector encoding the herpes simplex virus thymidine kinase (HSV-tk) gene. When combined with an oral antiviral prodrug (valacyclovir), this approach induces targeted tumor cell death and stimulates a systemic immune response. The study aims to characterize:

* Viral shedding and biodistribution of CAN-2409 genomes in blood, urine, and semen using validated qPCR assays.
* Immune activation biomarkers, including lymphocyte subsets, cytokine profiles, and circulating tumor-related proteins.

Approximately 30 patients with favorable risk prostate cancer and will receive 3 courses of injections of aglatimigene besadenovec followed by valacyclovir. EBRT will start after the second injection. Biospecimens (blood, urine, semen) will be collected before and after each injection to assess biodistribution and immune response.

Safety will be monitored continuously. Frequency of treatment-emergent adverse events (TEAEs) and laboratory values will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must give study-specific informed consent prior to enrollment
2. Histologically confirmed adenocarcinoma of the prostate
3. Participants meeting National Comprehensive Cancer Network (NCCN) favorable, intermediate-risk criteria
4. Participants must be planning and medically able to undergo standard or moderate hypofractionated prostate-only EBRT and able to tolerate multiple transrectal ultrasound guided injections
5. 18 years of age or older
6. Performance status must be Eastern Cooperative Oncology Group 0-2
7. The following laboratory criteria must be met:

   1. Aspartate aminotransferase (AST) < 3 x upper limit of normal
   2. Serum creatinine < 2 mg/dL
   3. Calculated creatinine clearance > 30 mL/min
   4. White blood cells > 3000/mm3
   5. Platelets >100,000/mm3

Exclusion Criteria:

1. Active liver disease, including known cirrhosis or active hepatitis
2. Participants on systemic corticosteroids (> 10 mg prednisone per day) or other immunosuppressive drugs
3. Known HIV+ participants
4. Regional lymph node involvement or distant metastases
5. Participants planning to receive whole pelvic irradiation
6. Other current malignancy (except squamous or basal cell skin cancers)
7. Other serious co-morbid illness or compromised organ function that, in the opinion of the Investigator, would interfere with treatment or follow-up. For example, participants with diseases that preclude radiation therapy to the prostate such as severe prostatitis and inflammatory bowel disease.
8. Prior treatment for prostate cancer except transurethral resection of the prostate (TURP). If prior TURP, participants must be deemed able to receive multiple intra-prostatic injections by the Investigator.
9. Participants who had or plan to have orchiectomy as the form of hormonal ablation
10. Known sensitivity or allergic reactions to acyclovir or valacyclovir

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of aglatimagene besadenovec | Up to 3 months post last injection of aglatimagene besadenovec.
  Evaluation of shedding of aglatimagene besadenovec viral genomes in urine, blood, and semen samples using validated bioassays over time.
Biomarkers of immune activation and tumor burden | Up to 3 months post last injection of aglatimagene besadenovec.
  Evaluation of prostate-specific antigen (PSA) ng/mL changes over time.
Biomarkers of immune activation and tumor burden | Up to 3 months post last injection of aglatimagene besadenovec.
  Evaluation of changes in lymphocytes as a proportion of total immune cells over time (lymphocytes/PBMCs).
Biomarkers of immune activation and tumor burden | Up to 3 months post last injection of aglatimagene besadenovec.
  Changes from baseline in concentrations of circulating proteins (e.g. Olink Normalized Protein Expression, or NPX).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Up to 3 months post last injection of aglatimagene besadenovec.
Treatment emergent toxicities in complete blood count, renal and hepatic clinical chemistries using CTCAE criteria | Up to 3 months post last injection of aglatimagene besadenovec.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Sheldon Freedman, MD Ltd., Las Vegas, Nevada
  - Summit Health, Saddle Brook, New Jersey